CLINICAL TRIAL: NCT03232671
Title: Role of Macrophage Migration Inhibitory Factor (MIF) in Heart Failure
Status: Completed | Type: Observational
Sponsor: University Hospital, Essen (Other)
Responsible Party: Principal Investigator, Fadi Al-Rashid, Dr., University Hospital, Essen
Other Study IDs: 15-6529-BO
Record Dates: First submitted 2017-07-25; First posted 2017-07-28 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Heart Diseases
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: MIF ELISA — Blood sample

SUMMARY:
Evaluating the additional value of Macrophage Migration Inhibitory factor (MIF) in cardiovascular diseases when assessed in clinical routine.

ELIGIBILITY:
Inclusion Criteria:

All patients presenting with symptoms of heart failure to the West-German Heart and Vascular Center according to the definition of the ESC 2016.

* Patients fulfilling criteria for the diagnosis of HFrEF
* Patients fulfilling criteria for the diagnosis of HFpEF
* Patients fulfilling criteria for the diagnosis of HFmrEF
* Patients presenting with dyspnea according to the NYHA classification I-IV, elevated BNP/NT-proBNP levels and echocardiographic findings of heart failure.

Exclusion Criteria:

* Age < 18 years
* Patients with symptoms of heart failure without fulfilling the criteria of the ESC guidelines 2016
* Denial to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients presenting with symptoms of heart failure.
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2020-04 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
180 days mortality | 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Peter Lüdike, M.D., Principal Investigator — University Hospital of Essen, Department of Cardiology and Vascular medicine
Locations (1):
- University Hospital of Essen, Essen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Luedike P, Alatzides G, Papathanasiou M, Heisler M, Pohl J, Lehmann N, Rassaf T. Predictive potential of macrophage migration inhibitory factor (MIF) in patients with heart failure with preserved ejection fraction (HFpEF). Eur J Med Res. 2018 May 4;23(1):22. doi: 10.1186/s40001-018-0321-1. PMID 29728137